CLINICAL TRIAL: NCT05925049
Title: An Observational Study Utilising Data From EU National MS Registries to Estimate the Incidence of Anti-Natalizumab Antibody Among Patients Who Receive Subcutaneous Administration of Natalizumab for Treatment of RRMS
Brief Title: A Study Utilising Data From European Union (EU) National Multiple Sclerosis (MS) Registries to Assess the Incidence of Anti-Natalizumab Antibody Among Participants Who Receive Subcutaneous Administration of Natalizumab for Treatment of Relapsing-remitting Multiple Sclerosis (RRMS)
Status: Active, not recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101MS412; EUPAS48753 (Other: EU PAS register number)
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Naive Participants: Per standard of care, participants with MS enrolled in selected MS registries, who are natalizumab-naïve and other MS mAb-therapy-naive will receive natalizumab 300 mg, SC injection according to decision of the treating physician.
  Interventions: Drug: Natalizumab
- Cohort 2: Natalizumab Experienced: Per standard of care, participants with MS enrolled in selected MS registries, who have previously received natalizumab IV will be switched from natalizumab IV to SC administration to receive natalizumab 300 mg, SC injection according to decision of the treating physician.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Administered as specified in the treatment arm.
  Other Names: Tysabri

SUMMARY:
The primary objective of this study is to estimate the incidence of Anti-Natalizumab Antibodies (ANAs) in the cohort of natalizumab-naïve and other MS monoclonal antibody (mAb)-naive participants who start receiving natalizumab subcutaneous (SC) injections. The secondary objectives of this study are to estimate the proportion of participants detected with ANAs when switched from natalizumab intravenous (IV) to natalizumab SC (natalizumab-experienced cohort); to evaluate serious adverse events (SAEs), including injection reactions and hypersensitivity reactions, by ANA status and to assess the proportion of participants who had MS relapse, by ANA status.

DETAILED DESCRIPTION:
The study will collect data prospectively and retrospectively.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who are natalizumab-naïve and other MS mAb-naive and who start on natalizumab SC.
* Participants who have previously received natalizumab IV and switch from natalizumab IV to SC administration.

Key Exclusion Criteria :

* For the natalizumab-naive and other MS mAb-naive cohort, participants who previously received natalizumab or other MS mAbs will be excluded.
* For the natalizumab-experienced cohort, participants who are naive to natalizumab will be excluded.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include available EU MS registry participants.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants in Natalizumab-Naive and Other MS mAb-Naive Cohort who Start Taking Natalizumab Injections and Develop Anti-Natalizumab Antibodies (ANAs) | Up to 1.75 years

SECONDARY OUTCOMES:
Percentage of Participants in Natalizumab-Experienced Cohort who Switched From Natalizumab IV Infusion to SC Injection and Develop Anti-Natalizumab Antibodies (ANAs) | Up to 1.75 years
Percentage of Participants With SAEs by Positive (Transient or Persistent) or Negative ANA Status | Up to 1.75 years
  SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in permanent or significant damage to health or limitation of capabilities or is manifested as a congenital anomaly or birth defect in offspring, irrespective of the administered dose of the medicinal product.
Percentage of Participants With MS Relapses by Positive (Transient or Persistent) or Negative ANA Status | Up to 1.75 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/